CLINICAL TRIAL: NCT04030416
Title: Clinical Accuracy Validation of the Medical Body Composition Analyzer Seca mBCA 555 in Comparison to Seca mBCA 515
Brief Title: Comparing Medical Body Composition Analyzer Seca mBCA 555 With Seca mBCA 515
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-21
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-10

CONDITIONS: Bioelectrical Impedance Measurement of Healthy Adults
Keywords: mBCA 555

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The mBCA 515 was compared to the gold standard methods MRI, DXA, ADP, D2O- and NaBr-dilution in previous clinical investigations (BCA-01, BCA-02, BCA-20) to generate prediction equations for calculating body composition (FFM, SMM, ECW, TBW and VAT) in different populations. Furthermore, normal ranges for body composition were generated based on the previous study BCA-03 conducted at the UKE.

The mBCA 555 is a new body composition analyzer measuring bioimpedance in standing position developed by seca.

In order to apply prediction equations and normal ranges from previous clinical investigations BCA-01, BCA-02, BCA-03 and BCA-20 to the new mBCA 555 it shall be compared to the mBCA 515.

DETAILED DESCRIPTION:
The use of bioelectrical impedance analysis (BIA) is widespread both in healthy subjects and patients. BIA allows the determination of the fat-free mass (FFM), skeletal muscle mass (SMM), fat mass (FM), extracellular water (ECW) and total body water (TBW) when using appropriate population, age or pathology-specific BIA equations and established procedures. BIA equations are based on validation studies where BIA is compared with reference methods such as Air Displacement Plethysmography (ADP), Dual-Energy X-Ray Absorptiometry (DXA), Magnetic Resonance Imaging (MRI) and isotope dilution.

The predicate device seca mBCA 515 was compared to the gold standard methods MRI, DXA, ADP, D2O- and NaBr-dilution in previous clinical investigations in Kiel (Germany) and New York City (USA) to generate prediction equations for calculating body composition (FFM, SMM, ECW, TBW and VAT) in different populations. Furthermore, normal ranges for body composition were generated in a previous study conducted at the University Hospital Hamburg-Eppendorf.

The mBCA 555 is a new body composition analyzer measuring bioimpedance in standing position developed by seca.

Primary objective is to test whether the mBCA 515 prediction equations can be applied to the new mBCA 555. If necessary, to proof substantial equivalence, prediction equations should be adjusted for the mBCA 555.

Secondary objective is to compare Impedance, phase angle, reactance and resistance for different frequencies in order to clarify if normal ranges for BIVA and phase angle generated with the mBCA 515 need to be adjusted for the new mBCA 555.

Bioimpedance was measured using the seca mBCA 555 and mBCA 515. Body height was measured using the seca 274.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects,
* 18 years and older,
* subjects need to be able to sign the informed consent and privacy policy

Exclusion Criteria:

* acute disease
* pregnancy
* intake of diuretics
* edema diagnosed by inspection and palpation of lower limbs
* paralysis e.g. after a stroke
* neurodegenerative diseases e.g. ALS
* tumors in treatment
* amputation
* electronic implants e.g. pacemaker
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the investigation site
* current alcohol abuse
* active prostheses
* electronic life-support systems, e.g. artificial heart, artificial lung
* portable electronic medical devices, e.g. ECG devices or infusion pumps
* metallic implants

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: healthy adults
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Peine, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf - Institute of Transfusion Medicine, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the blood donor service of the Institute of Transfusion Medicine. All subjects needed to be suitable for blood donation according to "Hämotherapie-Richtlinien nach §§ 12 a und 18 TFG", chapter 2.1.4. Blood donation was conducted after study examinations.
Groups:
- Healthy Blood Donors: single arm study with healthy blood donors
Period: Overall Study
Arm/Group | Healthy Blood Donors
Started | 120
Completed | 119
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: healthy male and female subjects 18years and older
  1 subject of the planed 120 subjects did not complete the study
Arm/Group | Healthy Blood Donors
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No valid measurement is available for ID 113, resulting in 119 valid measurements
  years | 40.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No valid measurement is available for ID 113, resulting in 119 valid measurements
  Participants
    Female | 57
    Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: No valid measurement is available for ID 113, resulting in 119 valid measurements
  Participants
    Hispanic or Latino | NA — not reported
    Not Hispanic or Latino | NA — not reported
    Unknown or Not Reported | 119
weight [Mean (Standard Deviation); unit: kg] — Population: No valid measurement is available for ID 113, resulting in 119 valid measurements
  kg | 78.0 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: SMM
Description: Skeletal muscle mass, bias of mBCA 555 in comparison to mBCA 515
Time Frame: 10min
Population: healthy blood donors
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Healthy Blood Donors
Number analyzed (Participants) | 119
kg | 0.34 (0.44)

2. Secondary Outcome: Phase Angle
Description: Phase angle at 50 kHz, bias of mBCA 555 in comparison to mBCA 515
Time Frame: 10 minutes
Population: healthy blood donors
Measure: Mean (Standard Error); unit: Degree
Arm/Group | Healthy Blood Donors
Number analyzed (Participants) | 119
Degree | 0.080 (0.079)

3. Other Pre Specified Outcome: R50RS
Description: resistance right body side, 50 kHz, bias of mBCA 555 in comparison to mBCA 515
Time Frame: 5 minutes
Measure: Least Squares Mean (Standard Deviation); unit: Ohm
Arm/Group | Healthy Blood Donors
Number analyzed (Participants) | 119
Ohm | -1.9 (5.15)

4. Other Pre Specified Outcome: R5RS
Description: resistance right body side, 5 kHz, bias of mBCA 555 in comparison to mBCA 515
Time Frame: 5 minutes
Measure: Least Squares Mean (Standard Deviation); unit: Ohm
Arm/Group | Healthy Blood Donors
Number analyzed (Participants) | 119
Ohm | -3.05 (6.12)

ADVERSE EVENTS:
Time Frame: 2 month
Description: No AE or SAE were observed
Groups:
- Single Arm Study: healthy blood donors
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04030416/Prot_SAP_000.pdf